CLINICAL TRIAL: NCT05439512
Title: Feasibility of Patient-specific Titanium Mesh Via A Transantral Approach for Repair of Orbital Floor Fractures.
Brief Title: Orbital Floor Fracture Repair by Titanium Mesh Via Transantral Approach.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aliaa Khalaf Abd Ellatief Mohamed, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3310
Record Dates: First submitted 2022-06-26; First posted 2022-06-30 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Orbital Fractures
MeSH Terms: conditions — Orbital Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- orbital floor fracture (Experimental): orbital floor fracture
  Interventions: Procedure: transantral orbital floor reconstruction by titanium mesh

INTERVENTIONS:
Procedure: transantral orbital floor reconstruction by titanium mesh — reconstruction of orbital floor fracture by patient specific titanium mesh
  Other Names: trans antral orbital floor reconstruction

SUMMARY:
The aim of the study is to evaluate the feasibility of CAD/CAM osteosynthesis mesh through a transantral surgical approach in the Repair of orbital floor fractures by means of clinical and radiographic findings.

DETAILED DESCRIPTION:
A CAD/CAM osteosynthesis mesh through a transantral approach should assumingly provide accurate reconstruction of the orbital volume and anatomy while eliminating the usual morbidity of lower eyelid approaches during orbital reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recent unilateral orbital floor fracture indicated for internal reconstruction -
* (isolated or in combination with other facial fractures)
* with existing or estimated enophthalmos based on radiographs and a contra-lateral healthy non-operated orbit.

Exclusion Criteria:

* Delayed cases (more than 2 weeks)
* previously operated cases
* bilateral orbital floor fracture.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
enophthamus | 6 months
  will calculate the amount of alteration and quantity of Enophthalmos by mean of a Post-Op Soft window CT scan in mm

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry,Cairo University, Cairo, Egypt